CLINICAL TRIAL: NCT07152288
Title: A Single-dose, Open-label, Phase I Study Comparing the Pharmacokinetics, Safety, and Pharmacodynamics of HSK39297 in Subjects With Mild and Moderate Hepatic Impairment and Normal Hepatic Function
Brief Title: Investigation of Pharmacokinetics,Safety,and Pharmacodynamics of HSK39297 in Subjects With Hepatic Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK39297-103
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): Subjects with mild hepatic impairment.
  Interventions: Drug: HSK39297 tablets
- Treatment group B (Experimental): Subjects with moderate hepatic impairment.
  Interventions: Drug: HSK39297 tablets
- Treatment group C (Experimental): Subjects with normal hepatic function
  Interventions: Drug: HSK39297 tablets

INTERVENTIONS:
Drug: HSK39297 tablets — oral
  Arms: Treatment group A
Drug: HSK39297 tablets — oral
  Arms: Treatment group B
Drug: HSK39297 tablets — oral
  Arms: Treatment group C

SUMMARY:
The study is being conducted to compare the pharmacokinetics, safety, and pharmacodynamics of HSK39297 in subjects with mild to moderate hepatic impairment and normal hepatic function

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the study procedures and methods, participate voluntarily and be able to complete the study according to the protocol requirements, and sign the informed consent form (ICF) in writing;
2. Aged 18-70 years old on the date of signing the ICF (including the threshold), both male and female;
3. At the time of screening, male subjects weighing no less than 50 kg and female subjects weighing no less than 45 kg; body mass index (BMI): 18~32 kg/m2 (including the threshold);
4. Normal or abnormal physical examination, 12-ECG, vital signs, chest frontal and lateral radiographs/CT, abdominal ultrasound, and laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function, etc.) in the screening and baseline periods were not clinically significant.
5. The demographic means of subjects in the normal liver function group (Group C) at screening must meet the following matching criteria:

   1. BMI matched to the hepatic impairment group (Group A + Group B) with a mean value ± 15%;
   2. Age-matched to the hepatic impairment group (Group A + Group B), mean ± 10 years;
   3. Sex-matched to liver impairment group (Group A + Group B), mean value ± 1 case;
6. Glomerular filtration rate (eGFR) ≥75 mL/min/1.73m2 calculated using the Chronic Kidney Disease Epidemiology Collaborative Study Group (CKD-EPI) formula;
7. Subjects with childbearing potential must agree to have no plans for childbearing and voluntarily use highly effective contraception with their partner from the time of signing the ICF until 1 month after administration of the test drug, and to avoid sperm/egg donation. Female subjects of childbearing potential must have a negative serum pregnancy test at both screening and baseline and not be breastfeeding.

   For subjects with hepatic impairment, the following inclusion criteria must also be met:
8. Not on medication within 4 weeks prior to screening, or have at least 4 weeks of stable medication for hepatic impairment and/or other co-morbidities requiring long-term treatment;
9. Child-Pugh classification of Class A or B (without the use of albumin within 14 days), which is chronic liver injury caused by previous primary liver diseases, including but not limited to non-alcoholic steatohepatitis, viral hepatitis (hepatitis B, hepatitis C), etc.

Exclusion Criteria:

1. Smoked an average of more than 5 cigarettes per day in the past 3 months or those who cannot comply with the prohibition of smoking during the trial;
2. Known or suspected (as judged by the researcher) immunodeficiency diseases or hereditary complement deficiencies;
3. Allergic to two or more allergens, or in the judgment of the investigator, may be allergic to the study drug or its components;
4. Screen those who have a history of heavy drinking in the past 3 months (with an average daily alcohol consumption of > 2 units of alcohol (1 unit = 285 mL of beer, or 30 mL of spirits, or 100 mL of wine)) or those with a positive breath alcohol test;
5. Disease or medical condition that, in the judgment of the investigator, may interfere with the absorption, distribution, metabolism, and excretion of the drug or that may reduce compliance;
6. History of capsular bacterial infection in the past; including but not limited to Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae type b, etc;
7. Severe trauma or undergone surgery within 2 weeks prior to screening, or plan to undergo surgery during the trial period;
8. Participated in a clinical trial of any other drug or medical device within 3 months prior to screening or plan to do so during the study period, or still within 5 half-lives of the drug prior to screening (whichever is longer);
9. A previous diagnosis of malignant tumors (excluding radically resected basal cell carcinoma of the skin, papillary thyroid carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix);
10. History of drug or substance abuse; or a positive urine drug test at screening;
11. Donated or lost ≥ 400 mL of blood within 30 days, or received a blood transfusion prior to screening;
12. QTcF (males) > 480 ms at screening, or other 12-ECG abnormalities judged by the investigator to be clinically significant or unsuitable for participation;
13. Difficulty in swallowing, collecting blood intravenously, or physically unable to tolerate blood collection, or not expected to complete the entire trial follow-up;
14. Vaccined within 2 weeks prior to dosing or plan to receive the vaccine during the study;
15. Positive result in the screening of any of the following indicators: hepatitis B surface antigen, hepatitis C antibody, HIV antibody, or syphilis antibody (hepatitis B surface antigen and hepatitis C antibody can be positive in subjects in the liver insufficiency group).
16. Any physical or psychological disease or condition that, in the judgment of the investigator, is likely to increase the risk of the trial, interfere with compliance with the protocol and ability to complete the trial.

    Additional exclusion criteria for subjects with hepatic impairment:
17. History of any serious disease other than the primary disease of the liver itself, or a history of and/or abnormal clinically significant clinical laboratory tests that, in the opinion of the investigator, may affect the results of the test, including, but not limited to, a history of circulatory, endocrine, neurological, gastrointestinal, urologic, or hematologic, immunologic, psychiatric, and metabolic disorders;
18. Liver failure, or cirrhosis with combination of hepatic encephalopathy (West-Haven Level 2 and above), hepatocellular carcinoma (except for those with Barcelona Clinic Liver Cancer (BCLC) stage 0 or those who have achieved radical treatment results), ruptured variceal hemorrhage of the esophagogastric fundus vein, and other complications that, in the judgment of the investigator, make the subject unsuitable for participation in the study;
19. On systemic hormones (except subjects on stable use of ≤ 5 mg/day of prednisone or equivalent doses of glucocorticoids) or other immunosuppressive agents within 4 weeks prior to screening, or more than 4 weeks from their last immunosuppressive therapy at screening but are still within the drug's efficacy period (as assessed by the investigator);
20. Alpha-fetoprotein > 20 ng/mL; hemoglobin (Hb) ≤ 70 g/L; alanine aminotransferase (ALT) or mentholatum aminotransferase (AST) ≥ 5 times the upper limit of normal (ULN); severe active bleeding or a platelet level ≤30×10⁹/L (except for those judged by the investigator to be in a stable state);
21. History of liver transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Cmax | Post-dose at day 1 to day 10.
  The maximum plasma concentration.
AUC0-t | Post-dose at day 1 to day 10
  Area under the concentration curve from time 0 to the last quantifiable concentration
AUC0-inf | Post-dose at day 1 to day 10
  Area under the concentration curve from time 0 to extrapolated infinite time

SECONDARY OUTCOMES:
Tmax | Post-dose at day 1 to day 10
  Time to maximum plasma concentration
t1/2 | Post-dose at day 1 to day 10
  Terminal half-life
CL/F | Post-dose at day 1 to day 10
  Apparent clearance
Vz/F | Post-dose at day 1 to day 10
  Apparent volume of distribution
Incidence and severity of adverse events | Screening period up to day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided